CLINICAL TRIAL: NCT00908635
Title: The Role of Angiopoietin, Angiopoietin Receptor Tie-2, and Vascular Endothelial Growth Factor in Sepsis-Induced Multi-Organ Dysfunction Syndrome
Brief Title: The Role of Angiopoietin, Tie-2, and Vascular Endothelial Growth Factor (VEGF) in Sepsis-Induced Multiple Organ Dysfunction Syndrome (MODS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Shu-Min Lin, Chang Gung Memorial Hospital
Other Study IDs: 96-1483B
Record Dates: First submitted 2009-05-25; First posted 2009-05-27 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Sepsis; Multiple Organ Dysfunction Syndrome
Keywords: sepsis; organ failure
MeSH Terms: conditions — Sepsis; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- survivor: survivors of patients
- fatalities: non-survivors of patients

SUMMARY:
This study is designated to determine serum concentrations of inflammatory mediators Ang-1, Ang-2, Ang-1/Ang-2 ratio, and Tie-2 in patients with sepsis-induced MODS and to investigate the association among increased permeability, inflammatory mediators, and these serum mediators in development of organ failure.

DETAILED DESCRIPTION:
Multiple Organ Dysfunction Syndrome (MODS) frequently leads to death in patients with sepsis. Our previous work has demonstrated that endothelial injury is closely associated with MODS development and mortality in septic patients. The sepsis-induced damage of endothelial cell membrane gives rise to increased capillary permeability. Evidence suggests that increased capillary permeability in patients with sepsis was associated with higher incidence of MODS and death during the ICU stay than those with decreased permeability. Angiopoietin (Ang) system is the key mediator for maintaining capillary permeability. Ang-2 triggers an inflammatory response and inducing permeability by activating the endothelium. In contrast, Ang-1 is anti-inflammatory, can inhibit adhesion molecule expression and attenuate permeability increase in different stimuli. The disrupted angiopoietin system has been reported in patients with sepsis, but the association between angiotension and MODS in septic patients has not been well addressed.

This study is designated to determine serum concentrations of Ang-1, Ang-2, Ang-1/Ang-2 ratio, and Tie-2 in patients with sepsis-induced MODS and to investigate the association among increased permeability, inflammatory mediators,autonomic dysfunction, and these serum mediators in development of organ failure. In addition, the study will incubate endothelial cells with septic patients' serum or tumor necrosis factor (TNF)-alfa, and determine the effects of ang-1 administration and blockade of ang-2 on disruption of endothelial cell structure, permeability increase, and expression of adhesion molecules. The study will also determine the signaling pathways and altered NF-kB dimmer composition that is responsible for the inhibitory effect for ang-1 administration on TNF-alfa-induced intercellular adhesion molecule (ICAM)-1 expression on endothelial surface.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have known origin of infection plus at least 2 of the following criteria of systemic inflammatory response syndrome:

  * fever > 38C or hypothermia < 36C;
  * heart rate > 90 beats/ minute;
  * respiratory rate > 20 breaths/minute or PaCO2< 32 mmHg or mechanical ventilation for an acute process;
  * WBC count > 12x109/L or < 4x109/L or > 10% immature neutrophils.

Exclusion Criteria:

* Age less than 18 years,
* Pregnant,
* Inability to provide informed, written consent,
* Patients with urologic trauma resulting in frank hematuria, urinary infection, or existing chronic renal disease (serum creatinine level > 2.0 mg/dL),
* Patients receiving nephrotoxic drugs, admitted to the hospital following a surgical procedure, or remaining in the ICU for < 72 hours will be also excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to ICU due to sepsis
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
mortality | in hospital mortality

SECONDARY OUTCOMES:
organ failure | In ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Min Lin, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Lin SM, Wang YM, Lin HC, Lee KY, Huang CD, Liu CY, Wang CH, Kuo HP. Serum thrombomodulin level relates to the clinical course of disseminated intravascular coagulation, multiorgan dysfunction syndrome, and mortality in patients with sepsis. Crit Care Med. 2008 Mar;36(3):683-9. doi: 10.1097/CCM.0B013E31816537D8. PMID 18431261